CLINICAL TRIAL: NCT06198192
Title: Effects of Pilates Exercises on Static and Dynamic Balance in Children With Hearing Impairment
Brief Title: Effects of Pilates Exercises on Hearing Impairment Children
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Riphah International University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: REC/RCR&AHS/23/0754
Record Dates: First submitted 2023-12-26; First posted 2024-01-10 (Actual); Last update posted 2024-06-13 (Actual); Status verified 2024-06

CONDITIONS: Hearing Impaired Children
Keywords: Balance; Hearing Impairment; Pilate exercises
MeSH Terms: conditions — Hearing Loss | interventions — Exercise Movement Techniques

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Balance Exercises (Active Comparator): This group will receive conventional exercises for balance.
  Interventions: Other: Conventional Therapy and Balance Exercises
- Pilates Exercises (Experimental): This group will receive Pilate exercises along with Balance exercises
  Interventions: Other: Pilates Exercises

INTERVENTIONS:
Other: Pilates Exercises — Ten repetitions of Pilates exercises will be performed with a 2-minute rest period between repetitions. Pilate group will receive the intervention program three times/week for total 10 weeks
  Arms: Pilates Exercises
Other: Conventional Therapy and Balance Exercises — this group receive conventional therapy along with balance exercises. Standing with feet together while the therapist sitting behind and manually locking the child knees, and then slowly tilt him to each side, forward and backward. Step standing with therapist behind the child guiding him to shift his weight forward then backward alternately. High step standing and try to keep balanced. Standing with manual locking of the knees then tries actively to stoop and recover. Equilibrium, righting and protective reactions training. Open environment gait training will be conducted with the different obstacles. Session includes three times/week for total 10 weeks
  Arms: Balance Exercises

SUMMARY:
This study will determine the effects of Pilates exercises on static and dynamic balance in children with hearing impairment. Children with hearing impairment often encounter challenges in their motor development, including difficulties in maintaining balance and mobility. Impaired balance and limited mobility can significantly impact their overall physical well-being and functional independence. Therefore, it becomes crucial to explore effective interventions that can address these specific needs and promote improve balance and mobility in this population. Pilates, a mind-body exercise approach, has gained recognition for its potential benefits in enhancing balance, flexibility, and core strength in various populations.

DETAILED DESCRIPTION:
A Randomized clinical trial will be conducted through convenient sampling. Subjects will randomly be allocated into two groups experimental group will receive balance exercises in addition to Pilate exercise while control group will receive will receive conventional therapy for strength, balance and postural stability. The duration of the treatment will be 10 weeks for 3 days a week for 45 minutes. Pediatric Balance Scale, Pediatric Reach Test (Pediatric Functional Reach Test) and Timed Up and Go Test will be used as outcome measure. Data will be analyzed on SPSS version 29.0; normality of the data will be checked and tests will be applied according to the normality of the data either it will be parametric test or non-parametric based on the normality.

ELIGIBILITY:
Inclusion Criteria.

* Age between 5 to10 years
* Having greater than 24 score of mini mental state examination (MMSE-C) for children
* Children diagnosed with congenital sensorIneural hearing impairment
* Having a hearing loss>75dB
* Able to follow instructions

Exclusion Criteria:

* Presence of any visual, physical or mental disability in addition to hearing loss, or any orthopedic or neurological problem that may affect balance
* Severe hearing losses were greater than75dB
* Parents or patient refuse to take part
* Have participated in other therapy programs during our intervention

Ages: 5 Years to 10 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 38 (Actual)
Dates: Start 2023-12-01 (Actual); Primary Completion 2024-02-05 (Actual); Study Completion 2024-02-05 (Actual)

PRIMARY OUTCOMES:
Pediatric Balance Scale | 10 weeks
  It is 14-item criterion-referenced measure that examines functional balance in the context of everyday tasks in the pediatric population in 3 domains sitting, standing and changing of position. It measures steady state and anticipatory balance activities of varying difficulty that will be performed with or without visual inputs. Item score from 0-4 which may be measured by the ability to perform the assessed activity. Item scores will be summed having maximum score of 56 points that indicate perfect score. Time of administration is 20 minutes. It has excellent test retest reliability in typically developmental child that is (ICC 0.850)
Pediatric Reach Test (Pediatric Functional Reach Test): | 10 weeks
  It is used to measure standing balance in pediatric population, it is only done in standing position. The standing position will be described first and target will be set under the supervision first forward reach will be tested and after this lateral reach will be tested. Reliability of this test is within rater (0.54, 0.88 ICC) and among the rater is (0.50, 0.93ICC)
Time Up and Go Test (TUG) | 10 weeks
  It provides valuable measures how quickly one can stand up, walk 10 feet, turn around, walk back and sit down. Patient sit in the chair on the command go patient rises from the chair walks 3 meters at comfortable and safe pace, turns, walk back to the chair and sits down. Timings begins with the instruction go and end when the patient is seated. Reliability of TUG test was high, with ICC of 0.99 for within-session reliability and 0.99 for test-retest reliability analyzes on CP children

CONTACTS AND LOCATIONS:
Overall Officials: Khushbakhat Butt, MS*, Principal Investigator — Riphah International University
Locations (1):
- Riphah International University, Lahore, Punjab Province, Pakistan

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Rajendran V, Roy FG. An overview of motor skill performance and balance in hearing impaired children. Ital J Pediatr. 2011 Jul 14;37:33. doi: 10.1186/1824-7288-37-33. PMID 21756300
- [Background] Melo RS, Lemos A, Paiva GS, Ithamar L, Lima MC, Eickmann SH, Ferraz KM, Belian RB. Vestibular rehabilitation exercises programs to improve the postural control, balance and gait of children with sensorineural hearing loss: A systematic review. Int J Pediatr Otorhinolaryngol. 2019 Dec;127:109650. doi: 10.1016/j.ijporl.2019.109650. Epub 2019 Aug 21. PMID 31466025